CLINICAL TRIAL: NCT00010920
Title: Preventing Cognitive Decline With Alternative Therapies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: P50AT000066-01P2 (NIH); P50AT000066-01 (NIH)
Record Dates: First submitted 2001-02-02; First posted 2001-02-05 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Dementia; Memory Disorders
MeSH Terms: conditions — Dementia; Memory Disorders | interventions — Ginkgo biloba extract

INTERVENTIONS:
Drug: Ginkgo Biloba Extract

SUMMARY:
Preventing dementia is an important goal for our aging population. This proposal is an initial 42 months study of the effect of standardized ginkgo biloba extract (GBE) on preventing or delaying cognitive decline in people age 85 years or older (the oldest old). The study focuses on the oldest old who present a distinct advantage for primary prevention studies because of their particularly high risk for developing mild cognitive impairment (MCI), a precursor to dementia. Because this is a population that has previously been out of the mainstream for use of alternative medicine, the safety of GBE in this age group will also be tested in this study. The study is randomized, placebo controlled and double blind. Approximately 200 elderly cognitively healthy subjects will be enrolled and followed for detection of conversion to MCI. This pilot study is viewed as a necessary first step in order to demonstrate that GBE, an alternative or complementary therapy, has a disease modifying effect on the brain, distinct from a symptomatic effect. The study will test the feasibility of the randomized start design, a trial design proposed as a method for discerning brain- or disease- modifying from symptomatic effects. The magnitude of biological effect of the treatments will also be assessed with volumetric quantitative MRI, a complementary means of confirming whether there is a brain modifying effect (measured as a decrease in brain volume loss with treatment). Peripheral markers of oxidation status will measure possible anti-oxidant effects of GBE.

DETAILED DESCRIPTION:
See brief summary

ELIGIBILITY:
Inclusion Criteria:

* Can identify a collateral informant who has frequent contact with the subject
* No memory complaints compared to others of same age group and has not sought attention for concerns about memory or cognition
* Normal memory function defined by an education-adjusted score on the Logical Memory Subscale of the Wechsler Memory Scale-Revised
* Mini-Mental State Examination Score >23
* Clinical Dementia Rating (CDR) of zero

Min Age: 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Dates: Start 1999-09; Study Completion 2004-12

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Jeffrey Kaye, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health Sciences University/Neurology, Portland, Oregon, United States